CLINICAL TRIAL: NCT04956237
Title: Retinal Surgery With or Without Anesthesiologist, Comparison of Surgeon and Patient's Comfort
Acronym: Retine-Foch
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_0138
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Retinal Disease
Keywords: Peribulbar surgery; Tenonian surgery; Retinal surgery; Surgeon comfort; Patient comfort
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tenonian surgery: Hospital recruitment with outpatient surgery without the presence of an anesthesiologist, without loco-regional anesthesia and without intravenous route
- Peribulbar surgery: Gold standard: City recruitment with outpatient surgery with the presence of an anesthesiologist and with loco-regional anesthesia

SUMMARY:
Retinal surgeries are now performed in some hospitals with sub-Tenon anesthesia to replace conventional peribulbar anesthesia. The advantages of performing the surgery with Tenonian anesthesia can be: the cost reduced due to the non-intervention of an anesthesiologist, no pre-operative anesthetic consultation, no waiting period for the effectiveness of the peribulbar anesthesia (15-20min to have the effect of anesthesia of the eye). In addition, there are more numerous and dangerous complications of peribulbar anesthesia than sub-Tenonian anesthesia, however it allows the eye to remain stationary and to perform precise surgery safely, as long as the patient does not move his head.

Performing a sub-Tenonian anesthesia also makes it possible to carry out surgeries more quickly, this method having an immediate effect and being performed by the surgeon, without the intervention of an anesthesiologist.

The edema effect under the post / conjunctiva swells the area around the eye and allows partial oculomotor limitation. Finally, for the patient, recovery is faster: no sedation or venous route.

To date, however, no study has proven that the surgeon can safely operate on the patient without increased complications compared to peribulbar anesthesia.

This study aims to show that simple sub-Tenonian anesthesia in a short outpatient circuit does not induce more pain or discomfort for the patient than a longer outpatient circuit with bed and anesthesiologist. No studies have been performed on purely local anesthesia without a venous route.

For this, patients operated on at the Foch hospital without an anesthesiologist under subtenon's anesthesia will be compared to patients operated on under peribulbar anesthesia with an anesthesiologist at the Pierre Cherest clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients with an indication for retinal surgery
* Not having opposed to participate in the study

Exclusion Criteria:

* Claustrophobia
* Unbalanced psychiatric pathology
* Inability to lie down
* Deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient over 18 years of age undergoing retinal surgery including retinal detachment, epi-retinal membrane-internal limiting peel, macular hole, implant dislocation, vitrectomy, revision of capsular rupture
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Comparison of the comfort and safety of the surgeon between patients operated with peribulbar or tenonian anesthesia | At the surgery
  Number of eye or head movements of the patient during the operation

SECONDARY OUTCOMES:
Comparison of the patient's comfort during the operation between the 2 groups | 15 minutes after the end of the surgery
  Postoperative Iowa Satisfaction with Anesthesia Scale (ISAS) Score rated from 11 (worse outcome) to 66 (better outcome)
Comparison of the patient's comfort during the operation between the 2 groups regarding pain | Preoperative, peroperative and 15 minutes post surgery
  Visual analogic scale (VAS) of pain during the surgery rated from 0 "No pain" to 10 "worst possible pain"
Comparison of operating time between the 2 groups | At the end of the surgery
  Operating time
Assessement of the security between the 2 groups | At the end of the surgery
  Intraoperative complications and peroperative events

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique Pierre Cherest, Neuilly-sur-Seine
  - Foch Hospital, Suresnes